CLINICAL TRIAL: NCT00152282
Title: A Phase II Pilot Study to Evaluate the Safety and Efficacy of J867 Administered With Estrogen to Postmenopausal Women
Brief Title: A Study to Evaluate the Safety and Effectiveness of Asoprisnil and Estrogen Administration to Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Cynthia Mattia-Goldberg, Abbott
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M00-198
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Amenorrhea; Postmenopause
Keywords: Postmenopausal; Amenorrhea; Hormone replacement therapy; HRT; asoprisnil
MeSH Terms: conditions — Amenorrhea | interventions — asoprisnil; Estrogens, Conjugated (USP)

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Asoprisnil/Premarin
- 2 (Experimental)
  Interventions: Drug: Asoprisnil/Premarin
- 3 (Experimental)
  Interventions: Drug: Asoprisnil/Premarin
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo and Premarin

INTERVENTIONS:
Drug: Asoprisnil/Premarin — Asoprisnil 5mg and Premarin 0.625 mg Tablets, oral Daily for 12 weeks
  Arms: 1
Drug: Asoprisnil/Premarin — Asoprisnil 10mg and Premarin 0.625 mg Tablets, oral Daily for 12 weeks
  Arms: 2
Drug: Asoprisnil/Premarin — Asoprisnil 25mg and Premarin 0.625 mg Tablets, oral Daily for 12 weeks
  Arms: 3
Drug: Placebo and Premarin — Placebo and Premarin 0.625 mg Tablets, oral Daily for 12 weeks
  Arms: 4

SUMMARY:
The objective of this study is to determine the safety and effectiveness of 3 asoprisnil doses when administered to postmenopausal women with Premarin® 0.625 mg.

DETAILED DESCRIPTION:
The objective of this study is to determine the safety and effectiveness of asoprisnil 5, 10, and 25 mg, compared to placebo, when administered to postmenopausal women, with Premarin® 0.625 mg, for 12 weeks. Pharmacodynamic effects to be assessed include bleeding pattern, endometrial biopsy results, and endometrial thickness. Safety assessments will include clinical laboratory results, physical examination with vital signs, pelvic and breast examinations, ultrasound results, and adverse events

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with an intact uterus
* Body mass index (BMI) between 18.0 - 33.0
* Good general health
* Endometrial thickness ≤ 4 mm by TVU
* No history or suspected endometrial hyperplasia
* Negative urine pregnancy test
* Pap smear in last 6 months with no evidence of malignancy or pre-malignant changes
* Mammogram without suspicion of malignancy within last 6 months
* Endometrial biopsy with no evidence of pathologic changes within last 6 months

Exclusion Criteria:

* Any abnormal lab result the study-doctor considers significant
* History of severe reaction to hormone therapy
* Receiving hormone therapy
* Currently using phytoestrogenic compounds, such as red clover, black cohosh (Promensil and Remifemin), dong quai, ginseng and soy isoflavones
* History or known or suspected cancer other than basal cell carcinoma
* Stenosis of the cervix
* History of reproductive endocrine disorder
* Washout requirement for hormonal therapy not met
* Ovarian mass
* Submucus or other symptomatic fibroid which would confound efficacy

Ages: 48 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2000-09; Primary Completion 2001-08 (Actual); Study Completion 2001-08 (Actual)

PRIMARY OUTCOMES:
Assessment of endometrium by endometrial biopsy | Week 12
Change from baseline in endometrial thickness as assessed by ultrasound | Week 12

SECONDARY OUTCOMES:
Frequency and amount of vaginal bleeding via patient diary. | Week 4, 8, and 12
Incidence of hot flushes | Week 4, 8, and 12
Presence or absence of endometrial hyperplasia. | Week 12
Response to global efficacy question regarding improvement in menopause symptoms. | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Abbott